CLINICAL TRIAL: NCT00954473
Title: Retrospective Study of Genetic Risk Factors for Osteosarcoma
Brief Title: Study of Blood Samples From Patients With Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AOST08B1; NCI-2011-02192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AOST08B1 (Other: Children's Oncology Group); AOST08B1 (Other: Children's Oncology Group); AOST08B1 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Localized Osteosarcoma; Metastatic Osteosarcoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-correlative (osteosarcoma genetic risk): Blood samples undergo polymorphism analysis of common single-nucleotide polymorphisms and haplotypes to examine genetic variation, gene-gene interactions, and the population structure.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies blood samples from patients with osteosarcoma. Studying the genes found in samples of blood from patients with osteosarcoma may help doctors identify biomarkers related to the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Conduct a large-scale candidate gene association study in osteosarcoma (OS) using cases from the national Children's Oncology Group (COG) OS biology study (P9851 and successor study AOST06B1).

SECONDARY OBJECTIVES:

I. Conduct a genome-wide association study (GWAS) of OS. II. Fine-map genomic regions associated with OS to identify putative functional loci.

III. Conduct whole-exome sequencing of germline OS deoxyribonucleic acid (DNA) samples.

IV. Investigate the functional implications of promising genetic variants associated with OS.

OUTLINE:

Blood samples undergo polymorphism analysis of common single-nucleotide polymorphisms and haplotypes to examine genetic variation, gene-gene interactions, and the population structure.

ELIGIBILITY:
Inclusion Criteria:

* Blood samples collected from clinical trials COG-P9851 and COG-AOST06B1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All osteosarcoma patients seen at COG institutions are eligible
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2009-01; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Hardy-Weinberg equilibrium on all SNPs | Baseline
  Determined on all SNPs by chi-square tests.
SNPs associated with OS | Baseline
  Logistic regression will be used to estimate odds ratios and 95% confidence intervals for the association between each SNP and OS under co-dominant, dominant and recessive genetic models. Stratified analyses will be conducted to examine sex, tumor subtype and outcome differences.
Gene-gene interactions | Baseline
  Assessed using a multiplicative model. Haplotypes will be constructed using both Bayesian and expectation-maximization algorithms. Differences between cases and controls will be evaluated with HaploStats which uses haplotype posterior probabilities as weights to update the regression coefficients in an iterative manner.
Survival outcomes | Baseline
  Kaplan-Meier survival curves will be used to determine outcome relative to genotype.
Whole-exome variant loci | Baseline
  Annotation and filtering of each whole-exome variant locus will be performed using a custom software pipeline. Variants in >= 2 OS cases will be validated, and then subsequently replicated in additional OS cases (samples previously received for the GWAS from international collaborators). Variants will also be evaluated for presence in known biologically plausible pathways and genes.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Savage, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States